CLINICAL TRIAL: NCT07313488
Title: Oxygen Saturation Monitoring During Transport Between the Operating Room and the Post-anesthesia Care Unit
Acronym: SpO2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9538
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Surgery
Keywords: Surgery; Oxygen saturation monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate whether continuous SpO₂ monitoring during transfer between the operating room and the Post-Anesthesia Care Unit (PACU) reduces the incidence of desaturations

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Patient scheduled for surgery under general anesthesia at the HUS between January 1, 2024 and April 30, 2025

Exclusion Criteria:

- Administration of premedication that may impair judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥ 18 years old) scheduled for surgery under general anesthesia at the HUS between January 1, 2024 and April 30, 2025
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of the incidence of desaturations | upon Arrival in the Recovery Room
  To evaluate whether continuous SpO₂ monitoring during transfer between the operating room and the PACU reduces the incidence of desaturations by recording:
  * The last SpO₂ reading taken upon leaving the operating room
  * The first SpO₂ reading taken upon arrival in the recovery room
  * The lowest SpO₂ reading taken during the transfer between the operating room and the recovery room (for patients monitored by pulse oximetry)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie - CHU de Strasbourg - France, Strasbourg, France